CLINICAL TRIAL: NCT02489578
Title: Management in Real-life of Patients Hospitalized With Community-acquired Pneumonia in China
Brief Title: A Retrospective Study on Hospitalized Patients With Community-acquired Pneumonia in China (CAP-China)
Acronym: RSCAP-China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Jishuitan Hospital (Other); Beijing Luhe Hospital (Other); Qingdao Municipal Hospital (Other); Qilu Hospital of Shandong University (Other); Beijing Huimin Hospital (Unknown); China-Japan Friendship Hospital (Other); Linzi Hospital (Unknown); Second Hospital of Beijing Armed Police Corps (Unknown); Kunming Yan'an Hospital (Unknown)
Responsible Party: Principal Investigator, Bin Cao, MD, Capital Medical University
Other Study IDs: NCT20150101
Record Dates: First submitted 2015-03-16; First posted 2015-07-03 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Community Acquired Pneumonia
Keywords: Community Acquired Pneumonia; health care associated pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: other — retrospective cohort study

SUMMARY:
The purpose of this study is to evaluate the disease burden of hospitalized patients with CAP and healthcare-associated pneumonia (HCAP) in real life of China .

DETAILED DESCRIPTION:
In China, the data about current management of patients hospitalized with CAP in the real-life setting is not available,type of pneumonia, selection of initial antibiotic, time to clinical stability, antibiotic choice anf modification,clinical outcomes and costs remain unclear.

In this study, we will collect comprehensive information on CAP and HCAP management patterns to evaluate the disease burden of hospitalized patients with CAP and HCAP in real life of China .to analyze microbiological characteristics,clinical manifestations,antibiotic regimens ,adherences to guidelines and effect on outcome in different groups of patients with CAP (> and = 65 years, different comorbidities ,risk factors) ,to investigate microbiological characteristics,clinical manifestations,antibiotic regimens ,adherences to guidelines and effect on outcome in different groups of disease severity with CAP ,to provide the difference on microbiological characteristics,clinical manifestations,antibiotic regimens ,and outcome between patients with CAP and HCAP ,to understand the current situation of antibiotic regimen ,to evaluate influence of different antibiotic regimens on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 14 years of age
* Patient meets the criteria of community acquired pneumonia
* Patient meets the criteria of healthcare-associated pneumonia

Exclusion Criteria:

* Patients <14 years of age
* Patient meets the criteria of hospital acquired pneumonia
* Known active tuberculosis or current treatment for tuberculosis
* Non-infectious pulmonary diseases
* HIV positive

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3000 patients with community acquired pneumonia who meet the below inclusion/ exclusion criteria will be recruited in China.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
treatment failure at 72h after initiation of antibiotics | Time from the first dose use of antibiotics to 72 hours
  treatment failure was defined as a change of antibiotics due to worsening signs or symptoms associated with pneumonia
in-hospital treatment failure due to multiple causes | Time from date of admission to discharge up to 1 week
  1)death in hospital;2)change of antibiotics due to worsening signs or symptoms of infection, 3) recurrence, defined as signs or symptoms of infection after completion of therapy requiring re-initiation of antibiotics

SECONDARY OUTCOMES:
Duration of intravenous antimicrobial therapy | 2 weeks
  Time from the first dose of intravenous antibiotics to date of stop of intravenous antibiotics ,participants will be followed for the duration of hospital stay
Hospital length of stay | 2 weeks
  Patients will be asked about hospitalization, date, Patients will be asked about hospitalization, date, participants will be asked about the time of admission and discharge
in-hospital mortality | 2 weeks
  Time from date of admission to date of discharge,participants will be followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, MD, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

REFERENCES:
- [Result] Yang SQ, Qu JX, Wang C, Yu XM, Liu YM, Cao B. Influenza pneumonia among adolescents and adults: a concurrent comparison between influenza A (H1N1) pdm09 and A (H3N2) in the post-pandemic period. Clin Respir J. 2014 Apr;8(2):185-91. doi: 10.1111/crj.12056. Epub 2013 Nov 26. PMID 24106842
- [Result] Cao B, Huang GH, Pu ZH, Qu JX, Yu XM, Zhu Z, Dong JP, Gao Y, Zhang YX, Li XH, Liu JH, Wang H, Xu Q, Li H, Xu W, Wang C. Emergence of community-acquired adenovirus type 55 as a cause of community-onset pneumonia. Chest. 2014 Jan;145(1):79-86. doi: 10.1378/chest.13-1186. PMID 24551881
- [Result] Qu J, Gu L, Wu J, Dong J, Pu Z, Gao Y, Hu M, Zhang Y, Gao F, Cao B, Wang C; Beijing Network for Adult Community-Acquired Pneumonia (BNACAP). Accuracy of IgM antibody testing, FQ-PCR and culture in laboratory diagnosis of acute infection by Mycoplasma pneumoniae in adults and adolescents with community-acquired pneumonia. BMC Infect Dis. 2013 Apr 11;13:172. doi: 10.1186/1471-2334-13-172. PMID 23578215
- [Derived] Han X, Wang H, Chen L, Wang Y, Li H, Zhou F, Xing X, Zhang C, Suo L, Wang J, Yu G, Wang G, Yao X, Yu H, Wang L, Liu M, Xue C, Liu B, Zhu X, Li Y, Xiao Y, Cui X, Li L, Liu X, Cao B. Impact of inhaled corticosteroid use on elderly chronic pulmonary disease patients with community acquired pneumonia. Chin Med J (Engl). 2024 Jan 20;137(2):241-243. doi: 10.1097/CM9.0000000000002936. Epub 2023 Dec 20. No abstract available. PMID 38111015
- [Derived] Han X, Liu X, Chen L, Wang Y, Li H, Zhou F, Xing X, Zhang C, Suo L, Wang J, Yu G, Wang G, Yao X, Yu H, Wang L, Liu M, Xue C, Liu B, Zhu X, Li Y, Xiao Y, Cui X, Li L, Cao B; CAP-China network. Disease burden and prognostic factors for clinical failure in elderly community acquired pneumonia patients. BMC Infect Dis. 2020 Sep 12;20(1):668. doi: 10.1186/s12879-020-05362-3. PMID 32919458
- [Derived] Han X, Zhou F, Li H, Xing X, Chen L, Wang Y, Zhang C, Liu X, Suo L, Wang J, Yu G, Wang G, Yao X, Yu H, Wang L, Liu M, Xue C, Liu B, Zhu X, Li Y, Xiao Y, Cui X, Li L, Purdy JE, Cao B; CAP-China network. Effects of age, comorbidity and adherence to current antimicrobial guidelines on mortality in hospitalized elderly patients with community-acquired pneumonia. BMC Infect Dis. 2018 Apr 24;18(1):192. doi: 10.1186/s12879-018-3098-5. PMID 29699493
- [Derived] Chen L, Zhou F, Li H, Xing X, Han X, Wang Y, Zhang C, Suo L, Wang J, Yu G, Wang G, Yao X, Yu H, Wang L, Liu M, Xue C, Liu B, Zhu X, Li Y, Xiao Y, Cui X, Li L, Uyeki TM, Wang C, Cao B; CAP-China network. Disease characteristics and management of hospitalised adolescents and adults with community-acquired pneumonia in China: a retrospective multicentre survey. BMJ Open. 2018 Feb 15;8(2):e018709. doi: 10.1136/bmjopen-2017-018709. PMID 29449294
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Influenza+pneumonia+among+adolescents+and+adults%3A+a+concurrent+comparison+between+influenza+A+(H1N1)+pdm09+and+A+(H3N2)+in+the+post-pandemic+period.
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Emergence+of+community-acquired+adenovirus+type+55+as+a+cause+of+community-onset+pneumonia
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Accuracy+of+IgM+antibody+testing%2C+FQ-PCR+and+culture+in+laboratory+diagnosis+of+acute+infection+by+Mycoplasma+pneumoniae+in+adults+and+adolescents+with+community-acquired+pneumonia.